CLINICAL TRIAL: NCT07076004
Title: Nourishing Hope: The Impact of Nutrition in Cancer Treatment and Recovery in Maine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Christine B. Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2000039692
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: Medically tailored grocery delivery; Diet Quality
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care Group with Delayed Medically Tailored Grocery Delivery (Active Comparator): Option to pick-up fresh produce (fruits and vegetables) once per week from clinic locations served by the Christine B. Foundation at any time during the six-month study. At the end of the six-month study, participants in this arm will receive a delivery of free medically tailored groceries each week for six-month. They can select preferred types of proteins, grains, fruits, and vegetables. The size of the grocery delivery is adjusted for the number of people living in the household.
  Interventions: Behavioral: Standard of Care Group with Delayed Medically Tailored Grocery Delivery
- Medically Tailored Grocery Group (Experimental): A delivery of free medically tailored groceries each week for the six-month study. They can select preferred types of proteins, grains, fruits, and vegetables. The size of the grocery delivery is adjusted for the number of people living in the household. They will also have the option to pick-up fresh produce (fruits and vegetables) once per week from clinic locations served by the Christine B. Foundation during the study.
  Interventions: Behavioral: Experimental: Medically Tailored Grocery Group
- Medically Tailored Grocery Plus Nutrition Counseling Group (Experimental): Delivery of free medically tailored groceries each week for the 6-month study. They can select preferred types of proteins, grains, fruits, and vegetables. The size of the grocery delivery is adjusted for the number of people living in the household. In addition to the grocery delivery, one of our Registered Dietitians will speak with these participants a total of 8 times during the 6-month study. These sessions with the dietitian can be done via telephone or videoconference (e.g., Zoom) and each session will last about 30 minutes. The sessions will occur in Week 1, Week 2, Week 4, Week 6, Week 9, Week 12, Week 16, and Week 20. These participants will also receive a free book that contains written information related to the counseling sessions as well as a recipe book. They will also have the option to pick-up fresh produce (fruits and vegetables) once per week from clinic locations served by the Christine B. Foundation during the study.
  Interventions: Behavioral: Medically Tailored Grocery Plus Nutrition Counseling Group

INTERVENTIONS:
Behavioral: Medically Tailored Grocery Plus Nutrition Counseling Group — Weekly delivery of medically tailored groceries plus 8 remote nutritional counselling sessions.
  Arms: Medically Tailored Grocery Plus Nutrition Counseling Group
Behavioral: Experimental: Medically Tailored Grocery Group — Weekly delivery of medically tailored groceries.
  Arms: Medically Tailored Grocery Group
Behavioral: Standard of Care Group with Delayed Medically Tailored Grocery Delivery — Option to pick up fresh produce weekly from participating clinics. Medically tailored grocery delivery will be available for 6 months beginning at the end of the study.
  Arms: Standard of Care Group with Delayed Medically Tailored Grocery Delivery

SUMMARY:
The primary objective of this study is to determine the effect of a 6-month pilot randomized controlled trial of medically tailored grocery delivery plus nutrition counseling vs. medically tailored grocery delivery alone vs. standard of care (with delayed grocery delivery alone) among 100 individuals with any stage and type cancer who reside in Maine on change in diet quality from baseline to 6-months.

The secondary objective is to assess the benefits of the intervention on change from baseline to 6-months on self-reported healthcare utilization (e.g., hospitalizations, emergency room visits), malnutrition, cancer-treatment related symptoms, food insecurity, quality of life, and financial toxicity. We will also evaluate feasibility and acceptability of the intervention in the target population.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effect of a 6-month intervention of medically tailored groceries plus nutrition counseling vs. medically tailored groceries alone vs. standard of care on diet and health outcomes among 100 cancer survivors who reside in Maine. This project will be conducted in partnership with the Christine B. Foundation which has been delivering medically tailored groceries to cancer survivors in Maine since 2020, but has not yet evaluated the impact of this nutrition program on important health outcomes in people living with cancer. The eligibility criteria matched the population of cancer survivors currently served by the Christine B. Foundation as we are testing the effect of their services on health-related outcomes in their target population. Given medically tailored meals and groceries have conferred health benefits in other patient populations, but there is limited research among cancer survivors, this highly innovative study and could provide evidence on the potential benefits of this type of nutrition intervention specifically for cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Ever been diagnosed with cancer
* Reside Hancock, Penobscot, Washington or Piscataquis county in Maine for the next 6 months

Exclusion Criteria:

* Seeing a dietitian regularly (at least once every two weeks)
* Planned long-term inpatient cancer treatment
* Receiving nutrition via IV also known as total parenteral nutrition
* Getting nutrition through a feeding tube
* Drinking more than 3 bottles of liquid meal replacements, such as Ensure, per day
* Received grocery delivery or grocery (not produce only) pick-up from the Christine B. Foundation in the past 3 months.
* Those with reduced mental capacity and unable to understand all the components of the study, including the details of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Diet Quality | Change from baseline to 6 months
  Recent diet will be assessed via food frequency questionnaire (FFQ). Diet quality will be calculated using the HEI-2020; range of 0 - 100, higher score indicating better diet quality.

SECONDARY OUTCOMES:
Food Insecurity | Change from baseline to 6 months
  United Stated Department of Agriculture 6-item questionnaire; range of 0-6, higher score indicating lower food security.
Health Related Quality of Life | Change from baseline to 6 months
  12-item Short Form Survey (SF-12) will be used to generate the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Using norm based scores, above 50 indicate a better-than-average health-related quality of life.
Cancer-Treatment Related Symptoms | Change from baseline to 6 months
  Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). Count of number of symptoms.
Healthcare Utilization | Number from baseline to 6 months
  Self-reported visits and admissions to emergency rooms, urgent care clinics, and in-patient facilities.
Malnutrition | Change from baseline to 6 months
  Patient-Generated Subjective Global Assessment (PG-SGA); range of 0-33, higher score indicating greater likelihood of malnutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Leah M Ferrucci, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Public Health, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No